CLINICAL TRIAL: NCT07051109
Title: Comparison of Postoperative Recovery Between Dual-channel Pump for Intravenous Patient-controlled Analgesia(IV-PCA) and Conventional Single-channel Pump After Laparoscopic Sleeve Gastrectomy: a Prospective Randomized Controlled Trial
Brief Title: Dual-chamber Patient-controlled Analgesia for Postoperative Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Park InSun, Principal investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B-2208-775-002
Record Dates: First submitted 2025-01-12; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Morbid Obesity; PCA; Analgesia; PONV
MeSH Terms: conditions — Obesity, Morbid; Agnosia; Postoperative Nausea and Vomiting | interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dual-chamber PCA (Experimental)
  Interventions: Device: multimodal analgesia via dual-chamber PCA
- single regimen PCA (Active Comparator)
  Interventions: Device: single regimen (only fentanyl)

INTERVENTIONS:
Device: multimodal analgesia via dual-chamber PCA — combination of fentanyl and ketorolac through dual-chamber PCA
  Arms: dual-chamber PCA
Device: single regimen (only fentanyl) — fentanyl only through dual-chamber PCA
  Arms: single regimen PCA

SUMMARY:
Postoperative nausea and vomiting (PONV) are the most common complications that can occur after general anesthesia. Postoperative use of opioids and morbid obesity have been reported as risk factors of PONV. In this study, the investigators aimed to compare the degree of postoperative side effects and pain control when an intravenous patient-controlled analgesia combining fentanyl and ketorolac via a dual-chamber device was provided to participants undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Morbidly obese patients undergoing laparoscopic sleeve gastrectomy experience a relatively high incidence of postoperative nausea and vomiting, but no effective treatment method has been established yet to prevent them. Through this study, the investigators can expect that if a dual-chamber patient-controlled analgesia device can provide effective analgesia while reducing the amount of opioid used, and thus reduce postoperative nausea and vomiting, it can have the effect of increasing the quality of recovery and satisfaction of participants who have undergone laparoscopic sleeve gastrectomy. Furthermore, this dual-chamber patient-controlled analgesia device can be applied to various surgeries and various patient groups who are at risk for postoperative nausea and vomiting, and it is expected that it can be adapted as one of the methods to prevent postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 19 to 65 years
* American Society of Anesthesiologists physical status (ASA class) 1 to 3
* Patients scheduled for laparoscopic sleeve gastrectomy under general anesthesia
* Patients requesting the use of IV-PCA after surgery

Exclusion Criteria:

* Patients with hypersensitivity to the drugs used in this study (Ketorolac, Fentanyl)
* Patients with alcohol or drug dependence, long-term use of opioids or analgesics
* Patients with liver disease or renal failure
* Patients with peptic ulcer, patients with gastrointestinal bleeding predisposition
* Patients with suspected cerebrovascular hemorrhage, organic disorders of the head related to increased intracranial pressure
* Patients with bronchial asthma or bronchospasm symptoms
* Patients with severe respiratory depression
* Nasal polyps, angioedema
* Patients with or history of convulsive disease
* Patients for whom the use of neuromuscular blocking agents is contraindicated

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
postoperative nausea and vomitting | postoperative 1 day
  The Quality of Recovery score 15

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyunggi-do, South Korea